CLINICAL TRIAL: NCT06970470
Title: Efficacy of Spinal Orthoses in Functional Mobility of Older Adults With Hyperkyphosis: Study Protocol for a Randomized Clinical Trial
Brief Title: Efficacy of Spinal Orthoses on Mobility in Older Adults With Hyperkyphosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Collaborators: Financiadora de Estudos e Projetos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 7.097.128
Record Dates: First submitted 2024-12-11; First posted 2025-05-14 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2024-06

CONDITIONS: Hyperkyphosis
Keywords: Older Adults; Spinal Orthoses; Biomechanics
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Triple-Adjustable Posture Corrector - Thoracic Spinal Orthosis (Mercur®, Brazil) (Experimental): This intervention involves the daily use of the Triple-Adjustable Posture Corrector, a thoracic spinal orthosis manufactured by Mercur® (Santa Cruz do Sul, Brazil). The orthosis is used for postural support in older adults with hyperkyphosis. Participants will wear the orthosis for at least four hours per day during waking hours, excluding aquatic activities, bathing, and sleeping.
  Interventions: Device: Triple-Adjustable Posture Corrector Manufacturer: Mercur®, Santa Cruz do Sul, Brazil
- Generation Dynamic Osteoporosis Brace. (Experimental): This intervention involves the daily use of the Generation Dynamic Osteoporosis Brace, a thoracic spinal orthosis manufactured by Bort® (Weinstadt, Germany). Participants will wear the orthosis for at least four hours per day during waking hours, excluding aquatic activities, bathing, and sleeping.
  Interventions: Device: Generation Dynamic Osteoporosis Brace Manufacturer: Bort®, Weinstadt, Germany
- No Intervention - Control Group (No Intervention): Participants in this group will not use any spinal orthosis during the study period but will undergo the same biomechanical and functional assessments as the intervention groups.

INTERVENTIONS:
Device: Triple-Adjustable Posture Corrector Manufacturer: Mercur®, Santa Cruz do Sul, Brazil — The Triple-Adjustable Posture Corrector is a thoracic spinal orthosis designed to provide biomechanical support and postural correction in individuals with excessive thoracic kyphosis. It consists of elastic and adjustable non-rigid bands positioned around the shoulders and thorax, allowing individualized tension regulation. The brace promotes scapular retraction and axial alignment by increasing proprioceptive feedback and limiting thoracic flexion.
  Participants randomized to this intervention will be instructed to wear the orthosis for a minimum of four consecutive hours per day, during waking hours, for 16 weeks. The orthosis is to be removed during bathing, aquatic activities, and sleep. Individualized fitting will be provided at baseline by trained personnel, following the manufacturer's guidelines. Adherence will be monitored through self-reported daily logbooks. Participants will be advised to report discomfort, adverse effects, or perceived benefits.
  The primary clinical obje
  Arms: Triple-Adjustable Posture Corrector - Thoracic Spinal Orthosis (Mercur®, Brazil)
Device: Generation Dynamic Osteoporosis Brace Manufacturer: Bort®, Weinstadt, Germany — The Generation Dynamic Osteoporosis Brace is a semi-rigid thoracic orthosis designed to stabilize the spine and counteract the progression of hyperkyphosis, especially in populations at risk for vertebral fragility. The brace is composed of lightweight, breathable material, with anterior and posterior structural support and adjustable tension straps. It is intended to reduce spinal flexion, improve sagittal alignment, and facilitate back extensor activation.
  Participants assigned to this group will wear the orthosis for a minimum of four hours daily during waking hours, excluding sleep and aquatic activities, over a 16-week period. The orthosis will be individually fitted at the initial session by a trained physical therapist, following manufacturer protocols to ensure comfort, stability, and effectiveness. Participants will receive a daily logbook to record usage duration, comfort level, and perceived effects. Adherence will be monitored weekly.
  The brace is intended to improve trun
  Arms: Generation Dynamic Osteoporosis Brace.

SUMMARY:
This study investigates whether wearing specific back braces (spinal orthoses) can improve movement and physical function in older adults (60 years and older) with hyperkyphosis, a forward curvature of the upper spine. By testing two types of braces, the study seeks to find effective ways to manage hyperkyphosis and enhance mobility, independence, and quality of life in this population.

Study Purpose

The purpose is to evaluate the impact of two types of thoracic spinal orthoses on functional mobility, which includes walking, muscle function, and overall physical activity. This information will help healthcare providers better understand how braces can be used to manage hyperkyphosis and improve daily functioning for older adults.

Who Can Participate?

The study will include adults aged 60 or older who have been diagnosed with hyperkyphosis. Eligible participants will be randomly assigned to one of three groups:

1. Group 1: Participants will use the Triple-Adjustable Posture Corrector (TAPC), a brace designed to improve posture and reduce kyphosis.
2. Group 2: Participants will use the Generation Dynamic Osteoporosis Brace (G-DOB), another type of spinal brace targeting posture and mobility.
3. Control Group: Participants will not wear any brace.

How the Study Works

The study will run for 16 weeks. Participants in the brace groups will wear their assigned braces throughout the day, except during specific activities like bathing, sleeping, and swimming. No other changes to their daily routines will be required.

At the start and end of the study, participants will undergo assessments to measure their physical function and mobility. These assessments will include:

* Gait analysis: Evaluates walking patterns using advanced 3D motion technology.
* Muscle strength and joint function testing: Measures how well muscles and joints are working using isokinetic dynamometry.
* Muscle activity recording: Tracks how muscles respond during movement using surface electromyography (EMG).
* Physical activity monitoring: Captures activity levels using accelerometers, which are small devices that track movement.

Why Is This Study Important?

Hyperkyphosis can lead to challenges in daily life, such as difficulty walking, decreased balance, pain, and a higher risk of falls. While physical therapy and exercise are common treatments, many older adults need additional support to manage the condition. Spinal orthoses may offer a practical, non-invasive option to improve posture, reduce symptoms, and increase physical activity.

By comparing the effects of these two braces, the study aims to:

1. Determine whether these orthoses improve functional mobility, such as walking and muscle performance.
2. Provide evidence to guide healthcare professionals in using braces to treat hyperkyphosis.
3. Develop a standardized approach for incorporating orthoses into the care of older adults with this condition.

Benefits for Participants

While the study focuses on research, participants may also experience direct benefits, such as:

* Improved posture and comfort while moving.
* Increased awareness of their physical health and function.
* Access to state-of-the-art assessments and expert support throughout the study.

How Will Results Be Used?

The findings will inform healthcare providers about the potential benefits of using spinal braces for older adults with hyperkyphosis. If successful, this research could lead to:

* Better treatment plans for patients.
* Increased availability of braces tailored for older adults.
* Improved quality of life for people living with hyperkyphosis.

Key Takeaways for Patients and Families

* Hyperkyphosis is a manageable condition, and this study explores a promising new way to support mobility and independence.
* Participation involves wearing a brace during regular daily activities and attending two comprehensive evaluations.
* The study is safe, non-invasive, and designed to minimize disruptions to daily life.

This research offers an exciting opportunity to improve care for older adults with hyperkyphosis. By understanding how braces affect movement and strength, healthcare providers can develop better tools and strategies to support aging populations. Families and caregivers can also benefit from knowing there are new, evidence-based options to help their loved ones stay active and independent.

DETAILED DESCRIPTION:
Objective: This study aims to present the protocol for evaluating the effects of spinal orthoses on the functional mobility of older adults with hyperkyphosis.

Design: This protocol outlines a randomized clinical trial with two intervention groups and one control group, to be conducted over 16 weeks. Participants will be older adults aged 60 years or older with a diagnosis of hyperkyphosis. They will be randomized to use one of two thoracic spinal orthoses (the Triple-Adjustable Posture Corrector or the Generation Dynamic Osteoporosis Brace). The intervention will involve continuous orthosis use, excluding aquatic activities, bathing, and sleep. Assessments will occur before and after the intervention period. Functional mobility will be measured through biomechanical parameters such as gait, joint torque, muscle activation, and physical activity levels, using 3D motion analysis, isokinetic dynamometry, surface electromyography, and accelerometry.

Conclusion: This study will evaluate the impact of spinal orthoses on the functional mobility of older adults with hyperkyphosis, enabling the development of a clinical application methodology for this population.

ELIGIBILITY:
Inclusion Criteria:

* Aged 60 years or older
* Clinical diagnosis of hyperkyphosis
* Ability to walk without assistive devices

Exclusion Criteria:

* Cognitive impairment
* Inability to complete the proposed assessments
* Non-compliance with orthosis use during the intervention period

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Thoracic Kyphosis Angle (degrees) | Baseline (Week 0) and post-intervention (Week 16)
  Thoracic spinal curvature will be assessed using the Goniometer-Pro® mobile application (Digiflex, USA), which provides a validated digital estimation of the Cobb angle in degrees. The measurement will be performed in the standing position with anatomical reference points on the thoracic spine. Two consistent measures will be averaged. This outcome evaluates structural postural changes over time.
Gait Speed (meters/second) | Baseline (Week 0) and post-intervention (Week 16)
  Walking speed will be measured in meters per second using the BTS SMART-D™ 3D motion capture system and a synchronized resistive pressure platform (PWalk 3000, BTS Engineering, Italy). Participants will walk at self-selected speed over a flat walkway, and the average of three valid trials will be reported.
Stride Length (centimeters) | Baseline (Week 0) and post-intervention (Week 16)
  Stride length will be assessed using the BTS SMART-D™ 3D motion capture system with markers placed according to the modified Helen Hayes protocol. The mean stride length from three valid gait trials will be calculated.
Step Width (centimeters) | Baseline (Week 0) and post-intervention (Week 16)
  Step width will be measured in centimeters using synchronized 3D motion capture and baropodometric analysis. The mediolateral distance between foot placements will be averaged from three valid walking trials.
Peak Plantar Pressure (kilopascals) | Baseline (Week 0) and post-intervention (Week 16)
  Peak plantar pressure will be recorded using the PWalk 3000 resistive pressure platform (BTS Engineering). Maximum pressure (kPa) detected during the stance phase of gait will be extracted and averaged across trials.
Support Phase Duration (milliseconds) | Baseline (Week 0) and post-intervention (Week 16)
  The duration of the support phase (ms) for each foot during gait will be measured using pressure platform data synchronized with 3D motion capture. The mean of three valid gait cycles will be used.
Trunk Muscle Torque (Newton-meters) | Baseline (Week 0) and post-intervention (Week 16)
  Concentric and eccentric peak torque of trunk flexor and extensor muscles will be measured in Newton-meters using the HUMAC NORM™ isokinetic dynamometer. Participants will perform five maximal effort repetitions per contraction mode, and peak torque values will be reported.
Shoulder Muscle Torque (Newton-meters) | Baseline (Week 0) and post-intervention (Week 16)
  Peak concentric and eccentric torque (Nm) of internal and external shoulder rotator muscles will be measured bilaterally using the HUMAC NORM™ dynamometer. The test will follow a standardized shoulder positioning protocol. The highest value among five trials will be recorded for each contraction type.
Electromyographic Activity (microvolts RMS) | Baseline (Week 0) and post-intervention (Week 16)
  Surface electromyography (sEMG) will be collected using the BTS FREEEMG™ system. RMS values (µV) of selected trunk (erector spinae, rectus abdominis, obliques) and shoulder muscles (infraspinatus, subscapularis, teres minor, etc.) will be recorded during isokinetic tests. Data acquisition follows SENIAM recommendations.
Physical Activity Level (milli-gravity units) | 7 consecutive days before baseline (Week -1 to 0) and after final intervention week (Week 15 to 16).
  Daily physical activity will be measured using ActiGraph™ GT3X accelerometers worn on the hip. The mean vector magnitude (mg) will be calculated from at least 4 valid days, excluding periods of sleep and aquatic activities.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael R Baptista, PhD, Principal Investigator — Pontifical Catholic University of Rio Grande do Sul
Locations (2):
- Brazil (2):
  - Pontifical Catholic University of Rio Grande do Sul., Porto Alegre, Rio Grande do Sul
  - Pontifical Catholic University of Rio Grande do Sul, Porto Alegre, Rio Grande do Sul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stegeman DF, Hermens HJ. Standards for surface electromyography: the European project "Surface EMG for non-invasive assessment of muscles (SENIAM)
- [Background] Yang S, Chen C, Du S, Tang Y, Li K, Yu X, Tan J, Zhang C, Rong Z, Xu J, Wu W, Luo F. Assessment of isokinetic trunk muscle strength and its association with health-related quality of life in patients with degenerative spinal deformity. BMC Musculoskelet Disord. 2020 Dec 9;21(1):827. doi: 10.1186/s12891-020-03844-8. PMID 33298028
- [Background] Dauty M, Delbrouck C, Huguet D, Rousseau B, Potiron-Josse M, Dubois C. Reproducibility of concentric and eccentric isokinetic strength of the shoulder rotators in normal subjects 40 to 55 years old. IES. 2003;11(2):95-100. doi:10.3233/IES-2003-0134
- [Background] Edouard P, Samozino P, Julia M, Gleizes Cervera S, Vanbiervliet W, Calmels P, Gremeaux V. Reliability of isokinetic assessment of shoulder-rotator strength: a systematic review of the effect of position. J Sport Rehabil. 2011 Aug;20(3):367-83. doi: 10.1123/jsr.20.3.367. PMID 21828388
- [Background] Valentini FA, Granger B, Hennebelle DS, Eythrib N, Robain G. Repeatability and variability of baropodometric and spatio-temporal gait parameters--results in healthy subjects and in stroke patients. Neurophysiol Clin. 2011 Oct;41(4):181-9. doi: 10.1016/j.neucli.2011.08.004. Epub 2011 Sep 13. PMID 22078730
- [Background] Kadaba MP, Ramakrishnan HK, Wootten ME, Gainey J, Gorton G, Cochran GV. Repeatability of kinematic, kinetic, and electromyographic data in normal adult gait. J Orthop Res. 1989;7(6):849-60. doi: 10.1002/jor.1100070611. PMID 2795325
- [Background] Sasaki J, Coutinho A, Santos C, et al. Orientações para utilização de acelerômetros no Brasil. Rev Bras Ativ Fís Saúde. 2017;22(2):110-126. doi:10.12820/rbafs.v.22n2p110-126
- [Background] Kochhann R, Varela JS, Lisboa CSM, Chaves MLF. The Mini Mental State Examination: Review of cutoff points adjusted for schooling in a large Southern Brazilian sample. Dement Neuropsychol. 2010 Jan-Mar;4(1):35-41. doi: 10.1590/S1980-57642010DN40100006. PMID 29213658
- [Background] Koele MC, Lems WF, Willems HC. The Clinical Relevance of Hyperkyphosis: A Narrative Review. Front Endocrinol (Lausanne). 2020 Jan 24;11:5. doi: 10.3389/fendo.2020.00005. eCollection 2020. PMID 32038498
- [Background] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880
- [Background] Serrao M, Casali C, Ranavolo A, Mari S, Conte C, Chini G, Leonardi L, Coppola G, DI Lorenzo C, Harfoush M, Padua L, Pierelli F. Use of dynamic movement orthoses to improve gait stability and trunk control in ataxic patients. Eur J Phys Rehabil Med. 2017 Oct;53(5):735-743. doi: 10.23736/S1973-9087.17.04480-X. Epub 2017 Jun 19. PMID 28627859
- [Background] Veiskarami M, Gholami M, Aboutorabi A, Ahmadi Bani M, Khamesi E. Motor Control Changes in Trunk Muscles after Using Anatomical Posture Control Orthosis in the Elderly Hyperkyphotic Subjects. JMR. Published online September 26, 2022. doi:10.18502/jmr.v16i4.10762
- [Background] Caetano GM, Santos Neto APD, Santos LSC, Fhon JRS. Risco de quedas e seus fatores associados na pessoa idosa hospitalizada. Rev bras geriatr gerontol. 2023;26:e230155. doi:10.1590/1981-22562023026.230155.pt
- [Background] Hosseinabadi M, Kamyab M, Azadinia F, Sarrafzadeh J. Effect of a Spinomed orthosis on balance performance, spinal alignment, joint position sense and back muscle endurance in elderly people with hyperkyphotic posture: A randomized controlled trial. Prosthet Orthot Int. 2020 Aug;44(4):234-244. doi: 10.1177/0309364620923816. Epub 2020 Jun 7. PMID 32507057
- [Background] Yao XM, Liu BB, Deng WY, Wang XH. The Awareness and Knowledge Regarding Sarcopenia among Healthcare Professionals: A Scoping Review. J Frailty Aging. 2022;11(3):274-280. doi: 10.14283/jfa.2022.7. PMID 35799432
- [Background] Seals DR, Justice JN, LaRocca TJ. Physiological geroscience: targeting function to increase healthspan and achieve optimal longevity. J Physiol. 2016 Apr 15;594(8):2001-24. doi: 10.1113/jphysiol.2014.282665. Epub 2015 Mar 11. PMID 25639909